CLINICAL TRIAL: NCT03034044
Title: POST-MARKETING SURVEILLANCE TO OBSERVE SAFETY AND EFFICACY OF XYNTHA SOLOFUSE PREFILLED SYRINGE
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1831086
Record Dates: First submitted 2016-11-30; First posted 2017-01-27 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2019-01

CONDITIONS: Factor VIII Deficiency, Congenital; Factor 8 Deficiency, Congenital; Autosomal Hemophilia A; Classic Hemophilia; Hemophilia A, Congenital
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
This study aims to observe the safety and efficacy of the Xyntha Solofuse prefilled syringe in the setting of routine practice. The primary objective is to detect medically significant events (factor VIII inhibitor). The secondary objective is to observe the overall efficacy and safety of the Xyntha Solofuse prefilled syringe including serious adverse events. In this open-label, non-comparative, observational, non-interventional, retrospective and multi-center study, post-marketing surveillance data will be collected retrospectively for up to 6 months from the initial administration day of the Xyntha Solofuse prefilled syringe injected into patients who have been administered the Xyntha Solofuse prefilled syringe.

As specified in the product approval issued by the Ministry of Food and Drug Safety, the study will be conducted for 4 years from the approval date. At least 600 study subjects will be enrolled in this study to meet the MFDS requirements. Although 600 is the assigned number of study subjects, the number of cases will be adjusted considering the actual number of enrolled subjects after the study start day.

ELIGIBILITY:
-. Inclusion criteria

To be eligible to enroll in this study, the study subjects will have to meet all the following inclusion criteria:

1. Hemophilia A (congenital factor VIII deficiency) patients who have been administered according to the indication of the product 1) Control and prevention of bleeding episodes and for routine and surgical prophylaxis in patients with hemophilia A (congenital factor VIII deficiency) 2) This drug does not contain von Willebrand factor and, therefore, is not indicated in von Willebrand's disease
2. Those who have been administered the Xyntha Solofuse prefilled syringe at least once - Exclusion criteria

Patients who satisfy the following criteria are not included in the study according to the local labeling:

1. Patients who have a history of hypersensitivity to the Xyntha Solofuse prefilled syringe or the ingredients of this drug.
2. Patients who have a history of hypersensitivity to hamster proteins.
3. Patients who have bleeding disorders other than hemophilia A.
4. Patients who have a history of FVIII inhibitors, or currently have or are suspected of having FVIII inhibitors. In case inhibitor titers quantified in Bethesda Units in the laboratory test results are within the normal laboratory range or at least 0.6 BU/mL. If laboratory tests cannot be performed, the investigator will determine whether or not inhibitors exist based on the clinical assessment results that show a decrease in efficacy of the replacement of FVIII (e.g. bleeding at least once, if the replacement of anti-bleeding agents is needed to be administered, and if frequency or dosage of replacement FVIII therapy needs to be increased).
5. Use of immunomodulatory therapy. (e.g. intravenous injection of immunoglobulin, use of regular systemic corticosteroids, cyclosporine, and mediators of anti-TNF-α)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is Hemophilia A (congenital factor VIII deficiency) patients who have been administered the Xyntha Solofuse prefilled syringe (as part of routine treatment at the Korean health care canter which has certified investigators).
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2018-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1831086&StudyName=Post+Marketing+Surveillance+To+Observe+Safety+And+Efficacy+Of+Xyntha+%28registered%29+Solofuse
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1831086&StudyName=Post-marketing+Surveillance+To+Observe+Safety+And+Efficacy+Of+Xyntha+Solofuse+Prefilled+Syringe

RESULTS

PARTICIPANT FLOW:
Groups:
- Xyntha: Participants who were prescribed with Xyntha Solofuse prefilled syringe, as part of routine treatment, were observed in this study for up to 6 months from the initial administration of Xyntha Solofuse.
Period: Overall Study
Arm/Group | Xyntha
Started | 106
Received Xyntha | 105
Completed | 105
Not Completed | 1
Not completed — Enrolled, but not received Xyntha | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all participants who received at least 1 dose of Xyntha solofuse prefilled syringe.
Arm/Group | Xyntha
Number analyzed (Participants) | 105
Age, Customized [Count of Participants; unit: Participants]
  < 30 years | 19
  30- 39 years | 29
  40- 49 years | 39
  50- 59 years | 11
  >= 60 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 105
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Race and Ethnicity were not collected from any participant. Population: Race and Ethnicity were not collected from any participant.
Duration of the disease, Continuous [Mean (Standard Deviation); unit: Years] — Duration of Hemophilia A in the study participants is provided in this baseline measure.
  Years | 32.4 (16.9)
Genetic mutation of factor VIII [Count of Participants; unit: Participants] — Presence of Genetic mutation of factor VIII was analyzed and provided in the categories of Yes (Present), No (not present) and Unknown.
  Participants
    Yes | 0
    No | 36
    Unknown | 69
Previous exposure to plasma-derived factor VIII [Count of Participants; unit: Participants] — Previous exposure of participants (before enrollment into the study) to plasma-derived factor VIII was determined and provided by using the categories as Yes (had exposure), No (did not have exposure) and Unknown.
  Participants
    Yes | 51
    No | 34
    Unknown | 20
Previous used factor VIII therapy [Count of Participants; unit: Participants] — Previous (before enrollment into the study) use of factor VIII therapy by participants was determined and provided by using the categories as Yes (had exposure) and No (did not have exposure).
  Participants
    Yes | 93
    No | 12
Personal history of allergic reactions to factor VIII products [Count of Participants; unit: Participants] — Personal history of allergic reactions to factor VIII products was analyzed and provided as in the categories of 'Yes' (had allergy) and 'No (did not have allergy)'.
  Participants
    Yes | 0
    No | 105
Family history of hemophilia A [Count of Participants; unit: Participants] — History of hemophilia A in the family of participants was determined and provided as in the categories of 'Yes' (had history of hemophilia disease) and 'No' (did not have history of hemophilia disease).
  Participants
    Yes | 23
    No | 82
Family history of factor VIII inhibitors [Count of Participants; unit: Participants] — History of factor VIII inhibitors in the family of participants was determined and provided as in the categories of 'Yes' (had history of factor VIII inhibitors) and 'No' (did not have history of factor VIII inhibitors).
  Participants
    Yes | 0
    No | 105
Family history of allergic reactions to factor VIII products [Count of Participants; unit: Participants] — History of allergic reactions to factor VIII products in the family of participants was determined and provided as in the categories of 'Yes' (had history of allergy) and 'No' (did not have allergy).
  Participants
    Yes | 0
    No | 105
Disease severity [Count of Participants; unit: Participants] — Disease Severity was determined based on activity of coagulation factor and was categorized into different level of categories which included as Mild (5 percent [%] to 40%), Moderate (1 to 5%) and Severe (less than [<] 1%).
  Participants
    Mild | 13
    Moderate | 8
    Severe | 80
    Unknown | 4
Medical history [Count of Participants; unit: Participants] — Medical history of hemophilia A in the family of participants was determined and provided as in the categories of 'Yes' (had history of hemophilia A) and 'No' (did not have history of hemophilia A).
  Participants
    Yes | 45
    No | 60
Renal Disorder [Count of Participants; unit: Participants] — Participants with renal disorder was determined and provided as in the categories of 'Yes' (had renal disorder besides Haemophilia A) and 'No'(did not have renal disorder).
  Participants
    Yes | 2
    No | 103
Hepatic Disorder [Count of Participants; unit: Participants] — Participants with hepatic disorder was determined and provided as in the categories of 'Yes' (had hepatic disorder besides Haemophilia A) and 'No' (did not have hepatic disorder).
  Participants
    Yes | 17
    No | 88
Personal History of Allergic Reactions to Factor VIII Products (within 12 months) [Count of Participants; unit: Participants] — Personal history of allergic reactions of participants to factor VIII products was analyzed and provided as in the categories of 'Yes' (had allergy) and 'No (did not had allergy)
  Participants
    Yes | 2
    No | 103
Concomitant treatments [Count of Participants; unit: Participants] — Concomitant treatments usage was determined in participants and provided here in the categories of 'Yes' (participants who had concomitant medication) and 'No (participants who did not have concomitant medication)'. Concomitant treatment included any other medicine/drug, which participants received other than Xyntha.
  Participants
    Yes | 36
    No | 69
Concomitant therapy [Count of Participants; unit: Participants] — Concomitant therapy was determined in participants and provided here in the categories of 'Yes' (participants who had receive concomitant therapy) and 'No (participants who did not have received concomitant therapy)'. Concomitant therapy included any other therapy which participants were received other than study therapy.
  Participants
    Yes | 2
    No | 103

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in participants who received Xyntha without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment Emergent Adverse Event (TEAE) was adverse event that started or worsened in severity after first administration of Xyntha Solofuse up to 6 months. AEs included both serious and non-serious adverse event.
Time Frame: From the first administration of Xyntha up to 6 months
Population: The safety population included all participants who received at least one dose of Xyntha Solofuse prefilled syringe.
Measure: Count of Participants; unit: Participants
Arm/Group | Xyntha
Number analyzed (Participants) | 105
Participants
  AEs | 15
  SAEs | 0

2. Primary Outcome: Number of Participants With Adverse Events (AEs) by Severity
Description: An AE was any untoward medical occurrence in participants who received Xyntha without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs were classified according to the severity in 3 categories a) mild - AEs does not interfere with participant's usual function b) moderate - AEs interferes to some extent with participant's usual function c) severe - AEs interferes significantly with participant's usual function, and was determined based on investigator's discretion.
Time Frame: From the first administration of Xyntha up to 6 months
Population: The safety population included all participants who received at least one dose of Xyntha Solofuse prefilled syringe. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Xyntha
Number analyzed (Participants) | 105
Participants
  Mild: number analyzed (Participants) | 15
  Mild | 10
  Moderate: number analyzed (Participants) | 15
  Moderate | 5
  Severe: number analyzed (Participants) | 15
  Severe | 0

3. Primary Outcome: Number of Participants Who Discontinued Due to Adverse Events
Description: An AE was any untoward medical occurrence in participants who received study drug without regard to possibility of causal relationship.
Time Frame: From the first administration of Xyntha up to 6 months
Population: The safety population included all participants who received at least one dose of Xyntha Solofuse prefilled syringe.
Measure: Count of Participants; unit: Participants
Arm/Group | Xyntha
Number analyzed (Participants) | 105
Participants | 0

4. Primary Outcome: Number of Participants With Treatment-Related Adverse Events (AEs) and Serious Adverse Events
Description: Treatment-related AE was any untoward medical occurrence attributed to Xyntha in a participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Relatedness to treatment was assessed by investigator. AEs included both serious and non-serious AEs.
Time Frame: From the first administration of Xyntha up to 6 months
Population: The safety population included all participants who received at least one dose of Xyntha Solofuse prefilled syringe.
Measure: Count of Participants; unit: Participants
Arm/Group | Xyntha
Number analyzed (Participants) | 105
Participants
  AEs | 2
  SAEs | 0

5. Primary Outcome: Number of Participants Who Died Due to Adverse Events
Description: An AE was any untoward medical occurrence in participants who received Xyntha without regard to possibility of causal relationship.
Time Frame: From the first administration of Xyntha up to 6 months
Population: The safety population included all participants who received at least one dose of Xyntha Solofuse prefilled syringe.
Measure: Count of Participants; unit: Participants
Arm/Group | Xyntha
Number analyzed (Participants) | 105
Participants | 0

6. Primary Outcome: Number of Participants With Overall Responses on a 4-Point Scale to the Injections Used to Treat Bleeding: On-Demand Treatment According to Surgery
Description: On-demand treatment according to surgery: treatment to increase factor in preparation for surgery. Overall responses to all injection of Xyntha Solofuse prefilled syringe used to treat bleeding in on-demand treatment (administration of an unscheduled dose of Xyntha Solofuse prefilled syringe to stop bleeding) according to surgery was assessed on 4 point scale of 1=excellent, 2=good, 3=moderate and 4=no response, higher score = better response. Excellent= Definite pain relief and/or improvement in signs of bleeding within 8 hours after an infusion, with no additional infusion, good= Definite pain relief and/or improvement in signs of bleeding within 8 hours after an infusion, with 1 additional infusion, moderate= Probable/slight improvement starting after 8 hours following infusion, with >=1 additional infusion administered for complete resolution of bleeding episode and no response= No improvement at all between infusions/during 24 hour interval following an infusion/condition worsens
Time Frame: From the first administration of Xyntha up to 6 months
Population: The efficacy analysis set included all participants who received at least one dose of Xyntha Solofuse prefilled syringe. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Xyntha
Number analyzed (Participants) | 6
Participants
  Excellent | 6
  Good | 0
  Moderate | 0
  No response | 0

7. Primary Outcome: Number of Participants With Overall Responses on a 4-Point Scale to the Injections Used to Treat Bleeding: On-Demand Treatment According to Bleeding
Description: On-demand treatment according to bleeding: treatment administered for spontaneous bleeding/abrasion; not requiring surgery. Overall responses to all injection of Xyntha used to treat bleeding in on-demand treatment (administration of an unscheduled dose of Xyntha Solofuse prefilled syringe to stop bleeding) according to bleeding was assessed on 4 point scale of 1=excellent, 2=good, 3=moderate,4=no response, higher score=better response. Excellent= Definite pain relief and/or improvement in signs of bleeding within 8 hours after an infusion, with no additional infusion, good= Definite pain relief and/or improvement in signs of bleeding within 8 hours after an infusion, with 1 additional infusion, moderate= Probable/slight improvement after 8 hours following infusion, with >=1 additional infusion administered for complete resolution of bleeding episode and no response= No improvement at all between infusions/during 24 hour interval following an infusion, or condition worsens.
Time Frame: From the first administration of Xyntha up to 6 months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Xyntha
Number analyzed (Participants) | 31
Participants
  Excellent | 28
  Good | 3
  Moderate | 0
  No response | 0

8. Primary Outcome: Number of Participants With Less Than Expected Therapeutic Effect (LETE): On-Demand Treatment According to Surgery
Description: LETE for on-demand treatment (administration of an unscheduled dose of Xyntha Solofuse prefilled syringe to stop bleeding) was defined as "no response" rated after each infusion of 2 consecutive infusions within 24 hours after on-demand treatment.
Time Frame: Within 24 hours of on-demand treatment (anytime within the observation period of 6 months)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Xyntha
Number analyzed (Participants) | 6
Participants | 0

9. Primary Outcome: Number of Participants With Less Than Expected Therapeutic Effect (LETE): On-Demand Treatment According to Bleeding
Description: LETE for on-demand treatment ((administration of an unscheduled dose of Xyntha Solofuse prefilled syringe to stop bleeding) was defined as "no response" rated after each infusion of 2 consecutive infusions within 24 hours after on-demand treatment) was defined as "no response" rated after each infusion of 2 consecutive infusions within 24 hours after on-demand treatment.
Time Frame: Within 24 hours of on-demand treatment (anytime within the observation period of up to 6 months)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Xyntha
Number analyzed (Participants) | 31
Participants | 0

10. Primary Outcome: Number of Infusions Required to Treat Each New Bleeding Episode
Description: It was calculated as total number of injections given throughout the study divided by total number of bleeding events.
Time Frame: From the first administration of Xyntha up to 6 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Infusions
Arm/Group | Xyntha
Number analyzed (Participants) | 31
Infusions | 1.22 (0.57)

11. Primary Outcome: Average Dose of Infusions Per Bleeding Event: On-Demand Treatment According to Surgery
Description: The average dose of Xyntha per bleeding event according to surgery in on-demand treatment was calculated as total dose of Xyntha (in IU) throughout the study divided by total number of bleeding event. On-demand treatment (administration of an unscheduled dose of Xyntha Solofuse prefilled syringe to stop bleeding) according to surgery means treatment to increase factor in preparation for surgery.
Time Frame: From the first administration of Xyntha up to 6 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: IU/event
Arm/Group | Xyntha
Number analyzed (Participants) | 6
IU/event | 2619.29 (1089.07)

12. Primary Outcome: Average Dose of Infusions Per Bleeding Event: On-Demand Treatment According to Bleeding
Description: The average dose of Xyntha per bleeding event was calculated as total dose of Xyntha throughout the study (in International Units [IU]) divided by total number of bleeding incidence. On-demand treatment (administration of an unscheduled dose of Xyntha Solofuse prefilled syringe to stop bleeding) according to bleeding means treatment administered due to spontaneous bleeding or abrasion.
Time Frame: From the first administration of Xyntha up to 6 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: IU/event
Arm/Group | Xyntha
Number analyzed (Participants) | 31
IU/event | 2140.08 (640.32)

13. Primary Outcome: Percentage of Participants With Bleeding Event
Time Frame: From the first administration of Xyntha up to 6 months
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Xyntha
Number analyzed (Participants) | 90
percentage of participants | 6.67

14. Primary Outcome: Annualized Bleeding Rates (ABRs)
Description: Annualized bleeding rate defined as number of bleeds under prophylactic setting (defined as bleeding occurred after 48 hours of prophylactic therapy [administration of Xyntha not for the treatment of a bleed but for the prevention of bleeding]) divided by (/) [(number of prophylactic therapy participants)*0.5)]
Time Frame: Within 48 hours after the prophylactic administration of Xyntha (within the duration of 6 months)
Population: as for outcome 6
Measure: Number; unit: bleeds per participant
Arm/Group | Xyntha
Number analyzed (Participants) | 90
bleeds per participant | 13.33

15. Primary Outcome: Number of Participants With Less Than Expected Therapeutic Effect (LETE): Prophylactic Therapy
Description: Less than expected therapeutic effect for prophylaxis therapy defined as breakthrough (spontaneous/non-traumatic) bleeding occurred within 48 hours of prophylaxis infusion (defined as: administration of Xyntha not for the treatment of a bleed but for the prevention of bleeding).
Time Frame: From the first administration of Xyntha up to 6 months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Xyntha
Number analyzed (Participants) | 90
Participants | 6

16. Primary Outcome: Average Dose of Infusions Per Bleeding Event: Prophylactic Therapy
Description: The average dose of Xyntha per bleeding event according to prophylaxis therapy treatment was calculated as total dose of Xyntha (in IU) throughout the study divided by total number of bleeding event. Prophylaxis therapy defined as breakthrough (spontaneous/non-traumatic) bleeding occurred within 48 hours of prophylaxis infusion (defined as administration of Xyntha not for the treatment of a bleed but for the prevention of bleeding).
Time Frame: From the first administration of Xyntha up to 6 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: IU/event
Arm/Group | Xyntha
Number analyzed (Participants) | 90
IU/event | 1881.33 (531.88)

17. Primary Outcome: Total Factor VIII Consumption
Description: Total factor VIII consumption for each participant was calculated by sum of the total amount of Xyntha Solofuse (in IU) infused for each Xyntha Solofuse infusion.
Time Frame: 6 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Xyntha
Number analyzed (Participants) | 90
IU | 106116.16 (55747.74)

ADVERSE EVENTS:
Time Frame: From the first administration of Xyntha Solofuse prefilled syringe up to 6 months
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis performed on safety analysis set.
Arm/Group | Xyntha
All-Cause Mortality (participants affected / at risk) | 22/105
Serious Adverse Events (participants affected / at risk) | 0/105
Other Adverse Events (participants affected / at risk) | 15/105
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xyntha (N=105)
Fever (General disorders) | 1
Hypertension (Cardiac disorders) | 2
Dizziness (Nervous system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 3
Factor VIII antibody positive (Vascular disorders) | 1
Haemorrhage NOS (Vascular disorders) | 1
Periodontal destruction (Gastrointestinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Skeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Sepsis (Infections and infestations) | 1
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 4
Haematuria (Renal and urinary disorders) | 1
Renal calculus (Renal and urinary disorders) | 1
Dermatitis fungal (Skin and subcutaneous tissue disorders) | 1
Laceration (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-05-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT03034044/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT03034044/SAP_001.pdf